CLINICAL TRIAL: NCT01750983
Title: A Phase I Trial of Ipilimumab (Anti CTLA- 4 Antibody) in Combination With Lenalidomide (IMiD) in Patients With Advanced Malignancies
Brief Title: Ipilimumab and Lenalidomide in Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0795; NCI-2013-00607 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Advanced Malignancies; Metastatic cancers; Ipilimumab; Yervoy; BMS-734016; MDX010; Lenalidomide; CC-5013; Revlimid
MeSH Terms: conditions — Neoplasms | interventions — Ipilimumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipilimumab + Lenalidomide (Experimental): Dose Escalation Group Ipilimumab Starting Dose: 1.5 mg by vein over 90 minutes on Day 1 of each 28 day cycle.
  Dose Escalation Group Lenalidomide Starting Dose: 10 mg by mouth on Days 1-21 of each 28 day cycle.
  Dose Expansion Group Starting Dose for Ipilimumab and Lenalidomide: Maximum tolerated dose (MTD) from Dose Escalation Groups.
  Interventions: Drug: Ipilimumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Ipilimumab — Dose Escalation Group Starting Dose: 1.5 mg by vein over 90 minutes on Day 1 of each 28 day cycle.
  Dose Expansion Group Starting Dose for Ipilimumab: Maximum tolerated dose (MTD) from Dose Escalation Group.
  Other Names: Yervoy; BMS-734016; MDX010
Drug: Lenalidomide — Dose Escalation Group Starting Dose: 10 mg by mouth on Days 1-21 of each 28 day cycle.
  Dose Expansion Group Starting Dose for Lenalidomide: Maximum tolerated dose (MTD) from Dose Escalation Group.
  Other Names: CC-5013; Revlimid

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of Yervoy® (ipilimumab) with Revlimid® (lenalidomide) that can be given to patients with advanced cancer. The safety of these drugs will also be studied.

Ipilimumab is designed to increase the immune system's ability to fight cancer.

Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. This may decrease the growth of cancer cells.

DETAILED DESCRIPTION:
Study Groups:

Dose escalation:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of the study drugs based on when you join the study.

Up to 5 dose levels of ipilimumab with lenalidomide will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of ipilimumab with lenalidomide is found.

Dose expansion:

Once the highest tolerable dose of ipilimumab with lenalidomide is found, up to 14 more participants may be enrolled. This will be to further study the safety of the combination of drugs at that dose and the level of effectiveness of the study drugs in a certain tumor group. This group will be called the dose expansion group.

Study Drug Administration:

Each study cycle is 28 days.

You will take lenalidomide by mouth on Days 1-21 of each cycle. You will swallow the capsules whole with water once a day. Do not break, chew, or open your capsules. The doctor will discuss this with you.

You will receive ipilimumab by vein over 90 minutes on Day 1 of each cycle. You will be monitored for side effects for 1-2 hours after the infusion.

Study Visits:

Every study visit:

° You will be asked if you have had any side effects.

Cycle 1:

* On Day 1: blood (about 4 teaspoons) will be drawn for routine tests.
* Between Days 2 and 7: If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.
* Between Days 8 and 14: Blood (about 4 teaspoons) will be drawn for routine tests. If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.
* Between Days 15 and 21: Blood (about 4 teaspoons) will be drawn for routine tests. If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.
* Between Days 22 and 28: Blood (about 4 teaspoons) will be drawn for routine tests. Your medical history will be recorded.

Cycle 2:

* On Day 1: Blood (about 4 teaspoons) will be drawn for routine tests.
* On Day 8 (+/- 3 days): Blood (about 4 teaspoons) will be drawn for routine tests.
* On Day 15 (+/- 3 days): Blood (about 4 teaspoons) will be drawn for routine tests.
* On Day 22 (+/- 3 days): Blood (about 4 teaspoons) will be drawn for routine tests.

Every other cycle (every 8 weeks):

° You will have an x-ray, CT scan, and/or PET/CT scan to check the status of the disease. ° Blood (about 1 tablespoon) will be drawn for tumor marker testing.

Before starting Cycle 3 and all following cycles:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any health problems you may have and any other drugs or herbal supplements you may be taking.
* Your performance status will be recorded.
* Blood (about 4 teaspoons) will be drawn for routine tests. Blood may be drawn more often if your doctor thinks it is needed.
* If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.

At the End of the study:

* Directly at the end of the study: If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.
* 28 days after therapy with lenalidomide stopped: If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.

Length of Dosing:

You may receive up to 4 doses of ipilimumab. You may continue receiving lenalidomide for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

You will be off study after your follow-up visit.

Follow-up:

You will have a follow-up-visit within 30 days after your last dose of study drugs. You will be asked about any health problems you may have and if you have had any side effects. If your study doctor thinks it is needed, you may have follow-up for a longer period of time. If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.

This is an investigational study. Ipilimumab is FDA approved and commercially available to treat metastatic melanoma. Lenalidomide is FDA approved and commercially available to treat multiple myeloma and myelodysplastic syndrome. Giving the combination of ipilimumab and lenalidomide to patients with advanced cancer is investigational.

Up to 101 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancers with no available standard therapy are eligible to enter the Phase 1 portion of this study.
2. Patients must be >/= 18 years.
3. Patients must be >/= 3 weeks beyond treatment with a cytotoxic chemotherapy regimen, or therapeutic radiation, or major surgery. A confirmation (written or verbal) that there is no risk of surgical complications from a patient's surgeon has to be obtained prior to starting therapy in patients with a history of major surgery within past 6 weeks. Patients may have received palliative localized radiation immediately before or during treatment provided that radiation is not delivered to the only site of disease being treated under this protocol. For biologic/targeted agents patients must be >/= 5 half-lives or >/= 3 weeks form the last dose (whichever comes first).
4. ECOG performance status </= 2.
5. Patients must have adequate organ and marrow function defined as: absolute neutrophil count >/= 1,000/mL platelets >/=50,000/mL; CrCl >/=60mL/min by Cockcroft -Gault calculation; total bilirubin </= 2x ULN (exceptions may apply to benign non-malignant indirect hyperbilirubinemia such as Gilbert syndrome); ALT(SGPT) </= 5X ULN; willingness to participate in the RevAssist® program. Females: two effective contraceptive methods should be used during therapy, during therapy interruptions, and for at least 4 weeks after completing therapy. Males: must always use a latex condom during any sexual contact with females of childbearing potential, even if they have undergone a successful vasectomy.
6. Patients must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

1. Uncontrolled intercurrent illness, including, but not limited to, uncontrolled infection, uncontrolled asthma, need for hemodialysis, need for ventilatory support.
2. Pregnant or lactating women.
3. History of hypersensitivity to ipilimumab.
4. History of hypersensitivity to lenalidomide.
5. Patients unwilling or unable to sign informed consent document.
6. Patients on hemodialysis.
7. History of organ transplantation.
8. History of autoimmune disease, including inflammatory bowel disease.
9. History of severe motor or sensory neuropathy, or any other autoimmune disorder which is deemed to be significant.
10. Patients with a prior history of Grade 4 rash associated with thalidomide treatment.
11. History of Angioedema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Ipilimumab in Combination With Lenalidomide | 28 days
  Maximum tolerated dose (MTD) defined as highest dose studied in which the incidence of dose limiting toxicity (DLT) was less than 33%.
Dose-Limiting Toxicities (DLT) of Ipilimumab in Combination With Lenalidomide | 28 days
  Dose-limiting toxicity (DLT) defined as any clinically grade 3 or 4 non-hematologic toxicity as defined in NCI CTC v4.0, expected and believed to be related to study medications (except nausea and vomiting, electrolyte imbalances responsive to appropriate regimens or alopecia), any grade 4 hematologic toxicity lasting at least 3 weeks or longer (as defined by the NCI-CTC v4.0) or associated with bleeding and/or sepsis; any grade 4 nausea or vomiting > 5 days despite maximum anti-nausea regimens, and any other grade 3 non-hematologic toxicity including symptoms/signs of vascular leak or cytokine release syndrome; or any severe or life-threatening complication or abnormality not defined in NCI-CTCAE v4.0 that is attributable to the therapy.

SECONDARY OUTCOMES:
Tumor Response | Every 8 weeks
  Rumor response defined as one or more of the following: (1) stable disease for more than or equal to 4 months, (2) decrease in measurable tumor (sentinel lesions) by more than or equal to 20% by RECIST criteria, (3) decrease in tumor markers by more than or equal to 25% (for example, a >/= 25% decrease in CA125 for patients with ovarian cancer), or (4) a partial response according to the Choi criteria

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org